CLINICAL TRIAL: NCT02523898
Title: Is the Co-administration of Metformine and CC as Compared to Placebo and CC Superior to Induce Ovulation in PCOS Patients With a Confirmed insulin-resistant-a Double Blind Randomized Clinical Trial
Brief Title: Metformine and CC Compared With Placebo and CC for Induction Ovulation in PCOS Patients With Insulin Resistant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unfortunately due to COVID 19and social problems following it,we were unable to reach the estimated sample size.Evantually we could have only 151 patients .
Sponsor: Semnan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Azam Azargoon, Director of Infertility ward., Semnan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SemnanUMS1
Record Dates: First submitted 2015-07-11; First posted 2015-08-14 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism
Keywords: Clomiphene; infertility; insuline resistant; metformine; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Infertility | interventions — Metformin; Sugars; Clomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformine and clomiphene citrate (Experimental): . metformin will be given at a dose of 500 mg three times a day for 8weeks. .In case of failure of ovulation after the end of this period, metformin was continued and patients were given 100 mg clomiphene for 5 days starting from day 3 of their spontaneous menses or withdrawal bleeding induced by progestin administration In cases of ovulation with CC without pregnancy, the patients were advised to participate in other two similar cycles of therapy with 100 mg clomiphene. When ovulation did not occur with 100 mg CC, its dose will be increased to 150 mg and the same treatment protocol will be used for this dose.
  Interventions: Drug: metformine; Drug: clomiphene citrate
- placebo and clomiphene citrate (Active Comparator): The patients in group two will be receiving placebo. In case of failure of ovulation after the end of this period, placebo was continued and patients were given 100 mg clomiphene for 5 days starting from day 3 of their spontaneous menses or withdrawal bleeding induced by progestin administration .In cases of ovulation with CC without pregnancy, the patients were advised to participate in other two similar cycles of therapy with 100 mg clomiphene.When ovulation did not occur with 100 mg CC, its dose will be increased to 150 mg and the same treatment protocol will be used for this dose. .
  10 days). .
  Interventions: Drug: placebo; Drug: clomiphene citrate

INTERVENTIONS:
Drug: metformine — 1500 mg metformine 8week plus 100 mg clomiphene for 5 days
  Other Names: Glucophage,Glumetza
  Arms: metformine and clomiphene citrate
Drug: placebo — placebo 8 weeks plus 100 mg clomiphene for 5 days
  Other Names: placebo,identical to metformine; sugar pill manufactured to mimic metformine 500mg
  Arms: placebo and clomiphene citrate
Drug: clomiphene citrate — 100 mg clomiphene for 5 days starting from day 3 of their spontaneous menses or withdrawal bleeding induced by progestin administration
  Other Names: clomid,serophene

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility which affects 12-21% of the population.Several studies performed evaluate the possible benefit of metformin alone or in combination with clomiphene (CC)as first-line treatment for infertility in women with PCOS have reported conflicting results. These conflicting results may be due to the presence or absence of insulin resistance(IR).Metformin decreases IR .However there is not a single randomized clinical trial with metformin in IR PCOS patients. Therefore, the aim of current study is to compare CC with coadministration of metformin and with CC with coadministration of placebo in IR PCOS patients to induce ovulation.

DETAILED DESCRIPTION:
Introduction:

PCOS is the most common cause of anovulatory infertility which affects 12-21% of the population. This percentage may vary according to the criteria used and population studied.Hyperandrogenism, chronic anovulation, and occasionally obesity are the characteristics of this syndrome. Currently, CC is the first-line infertility treatment in women with the PCOS .However, 20-25% of PCOS women fail to ovulate with incremental doses of CC and and do not respond due to resistance to CC .IR and hyperinsulinemia are considered as important factors in the pathogenesis of PCOS .Hence, lean and obese women with PCOS may have IR.Hyperinsulinism has been shown to play a part in ovarian hyperandrogenism and may directly influence and even prevent ovulation.Metformin, an insulin sensitizing agent, reduces levels of luteinizing hormone, hyperinsulinemia and also decreases ovarian production of androgens .For this reason a number of studies have been performed and evaluated the possible beneficial role of metformin in managing women with PCOS. However, the studies performed evaluate the possible benefit of metformin alone or in combination with CC as first-line treatment for infertility in women with PCOS have reported conflicting results .Recently a meta-analysis concluded that metformin was more burdensome than placebo, hence CC alone and not CC plus metformin should be the drug of choice in these patients.A high-quality Cochrane systematic review has reported on randomized controlled trials(RCTs) comparing metformin with CC in women with PCOS and demonstrated that CC had a significantly higher pregnancy and live birth rate in women with a BMI >30 kg/m2 whereas metformin had better results in women with a BMI <30 kg/m2.Lately, a meta-analysis reported that due to conflicting findings and heterogeneity across the included RCTs, there is insufficient evidence to establish a difference between metformin and CC in terms of ovulation, pregnancy, live birth, miscarriage and multiple pregnancy rates in nonobese women with PCOS. It was proposed that caution should be proceeded when prescribing metformin as first line pharmacological therapy in this group of women until further rigorous trials are done.

These conflicting results from the published studies may be due to the large differences and heterogeneity in study populations, particularly the possible presence or absence of IR. Metformin decreases IR, however there is not a single RCTwith metformin in IR PCOS patients. Therefore, the aim of current study is to compare CC with coadministration of metformin and with CC with coadministration of placebo in IR PCOS patients to induce ovulation.

Methods and materials:

A total of 388 IR women with PCOS will be enrolled in this study from infertility clinic at Amir-Al-Momenin Hospital, Semnan, Iran from november 2015 to april 2020 . All patients will be informed about the study and possible complications of the drugs by a consultant and informed consents will be signed. This study will be supervised and approved by the Research Council and Ethical Committee of Semnan University of Medical Sciences. For randomization random block allocation method was used, in which six blocks with four components will be present: AABB, BBAA, ABAB, BABA, ABBA, and BAAB. A random digit number table or generator to select and sort the blocks will be applied. The allocation sequence will be concealed in sequentially numbered, sealed envelopes.

This process will be prepared by a statistician from the Clinical Epidemiology Unit of Research Center. The corresponding envelope will be opened by a nurse who will be blinded to the study , after a patient was enrolled.

Sample size :

By taking the results of the study of Moll et al into account, which showed metformin plus CC resulted in 39.5 % pregnancy rate compared with 27.1% pregnancy rate with CC; and assuming that the results of the investigators' proposed study, which is done on IR women, are consistent with the results obtained from that study, the sample size calculated 388 by using the following formula, which compares the two proportions, and supposes the maximum error type 1 and 2 to be 5% and 20% respectively, provided that the two groups are equal and the trial is one sided.

Estimated sample size for two-sample comparison of proportions Test Ho: p1 = p2, where p1 is the proportion in population 1 and p2 is the proportion in population 2

Assumptions:

alpha = 0.0500 (one-sided) power = 0.8000 p1 = 0.3950 p2 = 0.2710 d=p1-p2=0.1240 n2/n1 = 1.00

Estimated required sample sizes:

n1 = 194 n2 = 194

Women will randomly be allocated to CC (100mg daily beginning on cycle day 3 for 5 days after spontaneous menses or withdrawal bleeding induced by progestin administration (medroxyprogesterone acetate [Provera], 5 mg per day for10 days and for up to 3 menstrual cycles.There is at least 5 days of pill free interval between progesterone(P) and clomid . The dose will be increased in subsequent cycles in cases of nonresponse (follicle <12mm by day 16 in CC cycle.) The maximum daily dose of clomiphene will be 150 mg (three pills), given for 5 days plus metformin (1500mgdaily has been starting before) (group A; n=194;) or CC plus placebo (group B; n=194).

Study Design:

All women will be examined clinically and their weight, height , body mass index (BMI) ,pulse and blood pressure will be recorded . These measurements will be taken by a nurse who will be unaware of the admission number of the patients. BMI will be calculated as weight divided by height squared (kg/m2). After an overnight fasting of 10 to 12 h, blood samples will be obtained for the determination of fasting blood glucose (FBG), insulin, FSH, LH, estradiol (E2), total and free testosterone (T), DHEAS, PRL, TSH, and 17OH progesterone for exclusion of 21-hydroxylasedeficient nonclassic adrenal hyperplasia (NCAH) on the 3rd day of a spontaneous menses or withdrawal bleeding induced by Provera.

All blood samples will be centrifuged and stored at -20°C until assayed together. Serum levels of FSH, LH, TSH and PRL will be measured using Enzyme-linked immunosorbent assay (ELISA,Wernecce,3200) (Ideal, Tehran, Iran). Total T, FreeT, DHEAS and insulin will be also measured using ELISA assay (Monobind,Inc,USA) . FBG will be measured using an enzymatic colorimetric method with Glucose Oxidase.Women with hypothyroidism included in this study after treatment and normal TSH(because in women with PCOS, a significant association between thyroid function, as reflected by TSH >2 mIU/l, and IR was found and the association appeared to be independent of age and BMI).

IR is determined with homeostatic model assessment( HOMA) method calculated by fasting insulin (mU/L) × fasting glucose (mmol/L)/ 22.5. The value of HOMA-IR ≥2.3 will be assumed as IR according to the Hosseinpanah et al studies´ in iranian women .After baseline studies are completed, the patients will be divided into two groups. In group1 metformin (Metformine, Chemidaro, Tehran, Iran) will be given at a dose of 500 mg three times a day for 8weeks. The dose will be increased from one to three tablets a day over a period of seven days to minimize side effects. The patients in group two will be receiving placebo (identical in appearance to metformin from the same factory).

The P levels in all subjects will be measured every other week in order to document ovulation. A P level > 5 ng/ml (16 nmol per liter) will considered as confirmatory of ovulation.

If pregnancy occurred, metformin will be continued for another 12 weeks. In case of failure of ovulation after the end of this period, metformin and placebo were continued and patients were given 100 mg CC (Clomid, Iran Hormone, Iran) for 5 days starting from day 3 of their spontaneous menses or withdrawal bleeding induced by Provera.Ovarian follicular response will be monitored by transvaginal sonography every other day from day 10 of the cycle by a single sonographist. When at least one follicle reached ≥18 mm in diameter, 5000 IU of HCG (Pregnyl; N.V. Organon, OSS, Netherlands) will be given intramuscularly and timed intercourse will advised (every other day for one week starting after receiving HCG). If there is no follicle ≥12mm by day 16 in CC cycle, the cycle will be presumed to be anovulatory and monitoring will be discontinued.

In cases of ovulation with CC without pregnancy, the patients will be advised to participate in other two similar cycles of therapy with 100 mg CC (group1 and 2). When ovulation will not occur with 100 mg CC, its dose will be increased to 150 mg and the same treatment protocol will be used for this dose. In group 1 metformine and in group 2 placebo will be continued through CC cycles.

Clinical pregnancy will be defined as the detection of at least one gestational sac on transvaginal ultrasound examination starting one week after the missed period.Ongoing pregnancy will be defined as the detection of fetal heart activity after 12 weeks of gestations.

Statistical analysis:

All the data will be entered to the SPSS software (Version 11.5.0, © SPSS Inc.), T-test (or Mann-Whitney test if needed),ANOVA for quantitative variables , Chi-square test and Fisher exact test if necessary for qualitative variables are used. P<0.05 will be considered significant in all tests.

ELIGIBILITY:
Inclusion Criteria:

* Insulin resistant ( HOMA-IR≥2.3) PCOS women between 20-36 years of age, with period of infertility more than 1 year and normal serum prolactin ,normal TSH after treatment , normal hystero salpingography and had no other infertility factor.

The diagnosis of PCOS according to the Rotterdam Criteria.

Exclusion Criteria:

* Diabetic women
* Any medication that could influence carbohydrate metabolism or pituitary-gonadal function at least 2 months before the study
* Hypertension or abnormal renal or liver function tests
* Ovarian drilling.

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 388 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
ovulation rate | every other weeks up to 8 weeks
  The progesterone levels will be measured every other week in order to document ovulation. A progesterone level > 5 ng/ml (16 nmol per liter) will considered as confirmatory of ovulation during metformine administration .Ovarian follicular response will be monitored by transvaginal sonography every other day from day 10 of the cycle to the 16th day of the cycle.ovulation will be confrmed When at least one follicle reached ≥18 mm in diameter.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 5 weeks of gestation
  Clinical pregnancy will be defined as the detection of at least one gestational sac on transvaginal ultrasound examination starting one week after the missed period
Ongoing pregnancy rate | 12 weeks of gestation
  Ongoing pregnancy will be defined as the detection of an alive fetus>12weeks of gestation on transvaginal ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Human M Fatemi, MD, Principal Investigator — Director GCC-Operations | Nova IVI Fertility LLC .Royale Marina Office, B22-23 P.O. 60202.Abu Dhabi/UAE; Azam Azargoon, MD, Principal Investigator — Abnormal Uterine Bleeding Research Center, Semnan University of Medical Sciences, Semnan, Iran.; Majid Mirmohammadkhani, Phd, Principal Investigator — Social Determinants of Health Research Center, Semnan University of Medical Sciences, Semnan, Iran.

REFERENCES:
- [Background] Franks S. Polycystic ovary syndrome. N Engl J Med. 1995 Sep 28;333(13):853-61. doi: 10.1056/NEJM199509283331307. No abstract available. PMID 7651477
- [Background] Moll E, van Wely M, Lambalk CB, Bossuyt PM, van der Veen F. Health-related quality of life in women with newly diagnosed polycystic ovary syndrome randomized between clomifene citrate plus metformin or clomifene citrate plus placebo. Hum Reprod. 2012 Nov;27(11):3273-8. doi: 10.1093/humrep/des310. Epub 2012 Aug 27. PMID 22926838
- [Background] Hammond MG. Monitoring techniques for improved pregnancy rates during clomiphene ovulation induction. Fertil Steril. 1984 Oct;42(4):499-509. doi: 10.1016/s0015-0282(16)48129-x. PMID 6436060
- [Background] Shepard MK, Balmaceda JP, Leija CG. Relationship of weight to successful induction of ovulation with clomiphene citrate. Fertil Steril. 1979 Dec;32(6):641-5. doi: 10.1016/s0015-0282(16)44411-0. PMID 510566
- [Background] Homburg R. Polycystic ovary syndrome. Best Pract Res Clin Obstet Gynaecol. 2008 Apr;22(2):261-74. doi: 10.1016/j.bpobgyn.2007.07.009. Epub 2007 Sep 5. PMID 17804299
- [Background] Chang RJ, Nakamura RM, Judd HL, Kaplan SA. Insulin resistance in nonobese patients with polycystic ovarian disease. J Clin Endocrinol Metab. 1983 Aug;57(2):356-9. doi: 10.1210/jcem-57-2-356. PMID 6223044
- [Background] Dunaif A, Graf M, Mandeli J, Laumas V, Dobrjansky A. Characterization of groups of hyperandrogenic women with acanthosis nigricans, impaired glucose tolerance, and/or hyperinsulinemia. J Clin Endocrinol Metab. 1987 Sep;65(3):499-507. doi: 10.1210/jcem-65-3-499. PMID 3305551
- [Background] Dunaif A, Segal KR, Futterweit W, Dobrjansky A. Profound peripheral insulin resistance, independent of obesity, in polycystic ovary syndrome. Diabetes. 1989 Sep;38(9):1165-74. doi: 10.2337/diab.38.9.1165. PMID 2670645
- [Background] Dunaif A, Segal KR, Shelley DR, Green G, Dobrjansky A, Licholai T. Evidence for distinctive and intrinsic defects in insulin action in polycystic ovary syndrome. Diabetes. 1992 Oct;41(10):1257-66. doi: 10.2337/diab.41.10.1257. PMID 1397698
- [Background] Nestler JE, Jakubowicz DJ, Evans WS, Pasquali R. Effects of metformin on spontaneous and clomiphene-induced ovulation in the polycystic ovary syndrome. N Engl J Med. 1998 Jun 25;338(26):1876-80. doi: 10.1056/NEJM199806253382603. PMID 9637806
- [Background] Nestler JE, Jakubowicz DJ. Lean women with polycystic ovary syndrome respond to insulin reduction with decreases in ovarian P450c17 alpha activity and serum androgens. J Clin Endocrinol Metab. 1997 Dec;82(12):4075-9. doi: 10.1210/jcem.82.12.4431. PMID 9398716
- [Background] Moll E, Bossuyt PM, Korevaar JC, Lambalk CB, van der Veen F. Effect of clomifene citrate plus metformin and clomifene citrate plus placebo on induction of ovulation in women with newly diagnosed polycystic ovary syndrome: randomised double blind clinical trial. BMJ. 2006 Jun 24;332(7556):1485. doi: 10.1136/bmj.38867.631551.55. Epub 2006 Jun 12. PMID 16769748
- [Background] Legro RS, Barnhart HX, Schlaff WD, Carr BR, Diamond MP, Carson SA, Steinkampf MP, Coutifaris C, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Giudice LC, Leppert PC, Myers ER; Cooperative Multicenter Reproductive Medicine Network. Clomiphene, metformin, or both for infertility in the polycystic ovary syndrome. N Engl J Med. 2007 Feb 8;356(6):551-66. doi: 10.1056/NEJMoa063971. PMID 17287476
- [Background] Sahin Y, Yirmibes U, Kelestimur F, Aygen E. The effects of metformin on insulin resistance, clomiphene-induced ovulation and pregnancy rates in women with polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2004 Apr 15;113(2):214-20. doi: 10.1016/j.ejogrb.2003.09.036. PMID 15063963
- [Background] Baran S, Api M, Goksedef BP, Cetin A. Comparison of metformin and clomiphene citrate therapy for induction of ovulation in the polycystic ovary syndrome. Arch Gynecol Obstet. 2010 Oct;282(4):439-43. doi: 10.1007/s00404-010-1497-y. Epub 2010 May 16. PMID 20473763
- [Background] Siebert TI, Viola MI, Steyn DW, Kruger TF. Is metformin indicated as primary ovulation induction agent in women with PCOS? A systematic review and meta-analysis. Gynecol Obstet Invest. 2012;73(4):304-13. doi: 10.1159/000335253. Epub 2012 Apr 17. PMID 22516925
- [Background] Jungheim ES, Odibo AO. Fertility treatment in women with polycystic ovary syndrome: a decision analysis of different oral ovulation induction agents. Fertil Steril. 2010 Dec;94(7):2659-64. doi: 10.1016/j.fertnstert.2010.03.077. Epub 2010 May 7. PMID 20451181
- [Background] Leanza V, Coco L, Grasso F, Leanza G, Zarbo G, Palumbo M. Ovulation induction with clomiphene citrate and metformin in women with polycystic ovary syndrome. Minerva Ginecol. 2014 Jun;66(3):299-301. PMID 24971785
- [Background] Xiao J, Chen S, Zhang C, Chang S. The effectiveness of metformin ovulation induction treatment in patients with PCOS: a systematic review and meta-analysis. Gynecol Endocrinol. 2012 Dec;28(12):956-60. doi: 10.3109/09513590.2012.705368. Epub 2012 Jul 19. PMID 22808990
- [Background] Tang T, Lord JM, Norman RJ, Yasmin E, Balen AH. Insulin-sensitising drugs (metformin, rosiglitazone, pioglitazone, D-chiro-inositol) for women with polycystic ovary syndrome, oligo amenorrhoea and subfertility. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD003053. doi: 10.1002/14651858.CD003053.pub4. PMID 20091537
- [Background] Misso ML, Costello MF, Garrubba M, Wong J, Hart R, Rombauts L, Melder AM, Norman RJ, Teede HJ. Metformin versus clomiphene citrate for infertility in non-obese women with polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2013 Jan-Feb;19(1):2-11. doi: 10.1093/humupd/dms036. Epub 2012 Sep 6. PMID 22956412
- [Background] Nawrocka-Rutkowska J, Ciecwiez S, Marciniak A, Brodowska A, Wisniewska B, Kotlega D, Starczewski A. Insulin resistance assessment in patients with polycystic ovary syndrome using different diagnostic criteria--impact of metformin treatment. Ann Agric Environ Med. 2013;20(3):528-32. PMID 24069859
- [Background] Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HW, Behre HM, Haugen TB, Kruger T, Wang C, Mbizvo MT, Vogelsong KM. World Health Organization reference values for human semen characteristics. Hum Reprod Update. 2010 May-Jun;16(3):231-45. doi: 10.1093/humupd/dmp048. Epub 2009 Nov 24. PMID 19934213
- [Background] Speroff L, Fritz MA. Induction ovulation In :Cilinical gynecologic endocrinology and infertility. 7th Ed. Philadelphi: Lippincott,Williams and Wilkins; 2005: 499-1180.
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Legro RS, Schlaff WD, Diamond MP, Coutifaris C, Casson PR, Brzyski RG, Christman GM, Trussell JC, Krawetz SA, Snyder PJ, Ohl D, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Santoro N, Eisenberg E, Zhang M, Zhang H; Reproductive Medicine Network. Total testosterone assays in women with polycystic ovary syndrome: precision and correlation with hirsutism. J Clin Endocrinol Metab. 2010 Dec;95(12):5305-13. doi: 10.1210/jc.2010-1123. Epub 2010 Sep 8. PMID 20826578
- [Background] Moll E, van der Veen F, van Wely M. The role of metformin in polycystic ovary syndrome: a systematic review. Hum Reprod Update. 2007 Nov-Dec;13(6):527-37. doi: 10.1093/humupd/dmm026. Epub 2007 Sep 1. PMID 17767003
- [Background] Karimzadeh MA, Javedani M. An assessment of lifestyle modification versus medical treatment with clomiphene citrate, metformin, and clomiphene citrate-metformin in patients with polycystic ovary syndrome. Fertil Steril. 2010 Jun;94(1):216-20. doi: 10.1016/j.fertnstert.2009.02.078. Epub 2009 May 21. PMID 19463994
- [Background] Parsanezhad ME, Alborzi S, Zarei A, Dehbashi S, Omrani G. Insulin resistance in clomiphene responders and non-responders with polycystic ovarian disease and therapeutic effects of metformin. Int J Gynaecol Obstet. 2001 Oct;75(1):43-50. doi: 10.1016/s0020-7292(01)00470-2. PMID 11597618
- [Background] Khorram O, Helliwell JP, Katz S, Bonpane CM, Jaramillo L. Two weeks of metformin improves clomiphene citrate-induced ovulation and metabolic profiles in women with polycystic ovary syndrome. Fertil Steril. 2006 May;85(5):1448-51. doi: 10.1016/j.fertnstert.2005.10.042. Epub 2006 Mar 31. PMID 16579997
- [Background] Legro RS, Brzyski RG, Diamond MP, Coutifaris C, Schlaff WD, Casson P, Christman GM, Huang H, Yan Q, Alvero R, Haisenleder DJ, Barnhart KT, Bates GW, Usadi R, Lucidi S, Baker V, Trussell JC, Krawetz SA, Snyder P, Ohl D, Santoro N, Eisenberg E, Zhang H; NICHD Reproductive Medicine Network. Letrozole versus clomiphene for infertility in the polycystic ovary syndrome. N Engl J Med. 2014 Jul 10;371(2):119-29. doi: 10.1056/NEJMoa1313517. PMID 25006718
- [Background] Hosseinpanah F, Barzin M, Tehrani FR, Azizi F. The lack of association between polycystic ovary syndrome and metabolic syndrome: Iranian PCOS prevalence study. Clin Endocrinol (Oxf). 2011 Nov;75(5):692-7. doi: 10.1111/j.1365-2265.2011.04113.x. PMID 21592169
- [Background] Hasegawa I, Murakawa H, Suzuki M, Yamamoto Y, Kurabayashi T, Tanaka K. Effect of troglitazone on endocrine and ovulatory performance in women with insulin resistance-related polycystic ovary syndrome. Fertil Steril. 1999 Feb;71(2):323-7. doi: 10.1016/s0015-0282(98)00454-3. PMID 9988406
- [Background] Johnson N. Metformin is a reasonable first-line treatment option for non-obese women with infertility related to anovulatory polycystic ovary syndrome--a meta-analysis of randomised trials. Aust N Z J Obstet Gynaecol. 2011 Apr;51(2):125-9. doi: 10.1111/j.1479-828X.2010.01274.x. Epub 2011 Jan 28. PMID 21466513
- [Background] Morin-Papunen L, Rantala AS, Unkila-Kallio L, Tiitinen A, Hippelainen M, Perheentupa A, Tinkanen H, Bloigu R, Puukka K, Ruokonen A, Tapanainen JS. Metformin improves pregnancy and live-birth rates in women with polycystic ovary syndrome (PCOS): a multicenter, double-blind, placebo-controlled randomized trial. J Clin Endocrinol Metab. 2012 May;97(5):1492-500. doi: 10.1210/jc.2011-3061. Epub 2012 Mar 14. PMID 22419702
- [Background] Lebovitz HE. Insulin resistance: definition and consequences. Exp Clin Endocrinol Diabetes. 2001;109 Suppl 2:S135-48. doi: 10.1055/s-2001-18576. PMID 11460565
- [Background] Palomba S, Falbo A, Orio F Jr, Manguso F, Russo T, Tolino A, Annamaria C, Dale B, Zullo F. A randomized controlled trial evaluating metformin pre-treatment and co-administration in non-obese insulin-resistant women with polycystic ovary syndrome treated with controlled ovarian stimulation plus timed intercourse or intrauterine insemination. Hum Reprod. 2005 Oct;20(10):2879-86. doi: 10.1093/humrep/dei130. Epub 2005 Jun 15. PMID 15958399
- [Background] DeUgarte CM, Bartolucci AA, Azziz R. Prevalence of insulin resistance in the polycystic ovary syndrome using the homeostasis model assessment. Fertil Steril. 2005 May;83(5):1454-60. doi: 10.1016/j.fertnstert.2004.11.070. PMID 15866584
- [Background] Goverde AJ, van Koert AJ, Eijkemans MJ, Knauff EA, Westerveld HE, Fauser BC, Broekmans FJ. Indicators for metabolic disturbances in anovulatory women with polycystic ovary syndrome diagnosed according to the Rotterdam consensus criteria. Hum Reprod. 2009 Mar;24(3):710-7. doi: 10.1093/humrep/den433. Epub 2008 Dec 17. PMID 19095675
- [Background] Mather K. Surrogate measures of insulin resistance: of rats, mice, and men. Am J Physiol Endocrinol Metab. 2009 Feb;296(2):E398-9. doi: 10.1152/ajpendo.90889.2008. No abstract available. PMID 19171846
- [Background] Wallace TM, Levy JC, Matthews DR. Use and abuse of HOMA modeling. Diabetes Care. 2004 Jun;27(6):1487-95. doi: 10.2337/diacare.27.6.1487. PMID 15161807
- [Background] Legro RS, Castracane VD, Kauffman RP. Detecting insulin resistance in polycystic ovary syndrome: purposes and pitfalls. Obstet Gynecol Surv. 2004 Feb;59(2):141-54. doi: 10.1097/01.OGX.0000109523.25076.E2. PMID 14752302
- [Background] Zheng J, Shan PF, Gu W. The efficacy of metformin in pregnant women with polycystic ovary syndrome: a meta-analysis of clinical trials. J Endocrinol Invest. 2013 Nov;36(10):797-802. doi: 10.3275/8932. Epub 2013 Apr 12. PMID 23580001
- [Background] Mueller A, Schofl C, Dittrich R, Cupisti S, Oppelt PG, Schild RL, Beckmann MW, Haberle L. Thyroid-stimulating hormone is associated with insulin resistance independently of body mass index and age in women with polycystic ovary syndrome. Hum Reprod. 2009 Nov;24(11):2924-30. doi: 10.1093/humrep/dep285. Epub 2009 Aug 3. PMID 19654109
- [Result] March WA, Moore VM, Willson KJ, Phillips DI, Norman RJ, Davies MJ. The prevalence of polycystic ovary syndrome in a community sample assessed under contrasting diagnostic criteria. Hum Reprod. 2010 Feb;25(2):544-51. doi: 10.1093/humrep/dep399. Epub 2009 Nov 12. PMID 19910321